CLINICAL TRIAL: NCT06823609
Title: A Phase I Clinical Study to Evaluate Safety, Tolerability, PK Characteristic and Preliminary Efficacy of QLS-1304 in Patients With Advanced Malignant Tumors
Brief Title: Phase I Clinical Study of QLS-1304 in the Treatment of Patients With Advanced Malignant Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Qilu Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: QLS1304-101
Record Dates: First submitted 2025-01-21; First posted 2025-02-12 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2025-01

CONDITIONS: Advanced Malignant Tumor

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- QLS1304 tablet (Experimental)
  Interventions: Drug: QLS1304 tablet

INTERVENTIONS:
Drug: QLS1304 tablet — QLS1304 monotherapy dose escalation and expansion

SUMMARY:
This study is a multi-center, open label, dose escalation/dose expansion phase I clinical trial aimed at evaluating the safety, tolerability, PK characteristics, and preliminary efficacy characteristics of QLS1304 monotherapy in patients with advanced malignant solid tumors. This study was divided into two stages: dose escalation and dose expansion.

ELIGIBILITY:
Inclusion Criteria:

* Volunteer to participate in this study, sign an informed consent form and have good compliance;
* Age ≥ 18 years old, Male or female
* ECOG score: 0-1
* Expected survival ≥ 12 weeks
* Local recurrent or metastatic advanced malignant solid tumor confirmed by histopathology or cytopathology;
* Failed to standard treatment or has no standard treatment scheme;
* Baseline presence of at least one evaluable lesion according to the RECIST v1.1;
* The functional level of important organs is basically normal, meeting the requirements of the scheme
* Female subjects with fertility and male subjects must agree to use highly effective contraception during the study treatment period and within 180 days after the last medication;
* Female subjects with fertility must have a negative serum HCG test within 7 days before the first medication in the study, and must be in non lactation.
* Volunteer to participate in this clinical trial, willing and able to follow the procedures related to clinical visits and research, understand the research procedures, and have signed informed consent

Exclusion Criteria:

* 1. Subjects have received live or attenuated live vaccines within 4 weeks before the first use of the investigational drug.
* Subjects have undergone major organ surgery within 4 weeks before the first use of the investigational drug.
* Subjects require long-term or high-dose use of non-steroidal drugs.
* Subjects have not recovered from adverse events (AEs) caused by previous anti-tumor treatment to ≤ grade 1.
* Subjects have a known or suspected severe allergy to theinvestigational drug or any of its components Subjects have other active malignant tumors within 5 years before the first use of the investigational drug.
* Subjects have brain metastases and/or carcinomatous meningitis or leptomeningeal disease.
* Subjects have active tuberculosis, radiation pneumonitis, drug-induced pneumonitis, pulmonary fibrosis, or other diseases, symptoms, or signs of severe lung function impairment.
* Subjects are unable to swallow tablets or had gastrointestinal abnormalities that the investigator assessed as potentially affecting drug absorption.
* Subjects have a history of severe cardiovascular or cerebrovascular disease within 6 months before the first use of the investigational drug.
* Subjects have a hypertension medial history that blood is not well controlled despite treatment with multiple antihypertension drugs.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2025-03-06 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Dose limited toxicity (DLT) of QLS1304 | up to 35 days
Maximum tolerated dose（MTD）of QLS1304 | up to 35 days
Recommended Phase II Dose (RP2D) of QLS1304 | up to 35 days

SECONDARY OUTCOMES:
adverse event | from the first drug administration to within 30 days for the last treatment dose
Cmax | through study completion, an average of 2 year
objective response rate(ORR) | through study completion, assessed up to 24 months
Tmax | through study completion, an average of 2 year
AUC0-t | through study completion, an average of 2 year
AUC0-inf | through study completion, an average of 2 year
CL/F | through study completion, an average of 2 year
Vd/F | through study completion, an average of 2 year
MRT | through study completion, an average of 2 year
t1/2 | through study completion, an average of 2 year

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Cancer Hospital, Shanghai, China